CLINICAL TRIAL: NCT06169618
Title: The Relationship Between Cervical Radiculopathy and Eye-hand Coordination
Acronym: CR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Saeed Ibrahim el Gabry, principle investigator Basma saeed ibrahim el gabry, Cairo University
Other Study IDs: P.T.REC/012/004095
Record Dates: First submitted 2023-11-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cervical Radiculopathy
Keywords: eye hand co ordination; cervical radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cervical radiculopathy group: thirty participants with cervical radiculopathy due to discogenic lesions.
  Interventions: Other: cervical radiculopathy
- normal group: thirty participants in normal without any discogenic lesion
  Interventions: Other: normal group

INTERVENTIONS:
Other: cervical radiculopathy — this group will have patients with cervical radiculopathy
  Groups: cervical radiculopathy group
Other: normal group — this group will have normal subjects
  Groups: normal group

SUMMARY:
this study will be conducted to investigate if there is a relationship between cervical radiculopathy and eye-hand coordination.

DETAILED DESCRIPTION:
Cervical radiculopathy is a disorder involving dysfunction of the cervical nerve roots commonly secondary to cervical spine degenerative changes such as disk herniation and/or foraminal stenosis compressing the nerve roots. Clinical manifestations are pain in neck and one or both of the upper extremities, as a result of compression or irritation of nerve roots in the cervical spine. It can be accompanied by motor, sensory, or reflex deficits. It is most common in persons 45-60 years of age, which result in terrible chronic pain. Eye hand coordination is the ability to do activities which require the simultaneous use of hands and eyes. It is a complex cognitive skill which unites visual and motor skills in the person and allowing the hands to guide by the visual stimulations. It lies at the core of our daily activities and interactions with objects and people around us as to be a defining characteristic of typical human life. Previous studies show that there was a marked alteration in the hand function in subjects with the cervical radiating pain. Since there was no study which investigated the relationship between cervical radiculopathy and eye hand coordination despite it is an important skill that adults use in countless activities of daily living and during working.

ELIGIBILITY:
Inclusion Criteria:

* Subjects normal with no neck complain.
* Patients of cervical radiculopathy due to cervical discogenic lesion.
* Ages range from 30-50 both males and females.
* Subjects should be able to follow simple verbal commands or instructions included in the procedures.

Exclusion Criteria:

* Participants with any neck trauma.
* Cervical Post-operative patients.
* Participants with vision deficiency.
* Participants with perceptual and cognitive problems with score less than 24 in mini mental state scale (Appendix I) (Goudsmit et al., 2018).
* Participants with any other neurological or musculoskeletal problems.
* Participants take medications that affect their attention.
* Participants have space-occupying lesions eg. tumors

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the first population will be thirty with cervical radiculopathy, the second group will be thirty subjects with the normal state
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
eye hand coordination movement speed objectively | baseline
  The Purdue Pegboard test will be used to assess eye hand coordination speed by putting as many pins as possible into the pegboard in 30 sec. the Test will be done three times each and averaged. The score for each of the four subtests
pain intensity | baseline
  numerical pain rating scale will be used for assessment of pain intensity. It is a single 11-point numeric scale. The physical therapist will ask the patient to state a number from 1 to 10 that best represents their perceived current pain intensity or pain intensity "in the last 24 hours". Zero usually represents 'no pain at all' whereas 10 is the upper limit represents 'the worst pain ever possible'
eye hand coordination accuracy and timing | baseline
  talking pen test will used to assess the accuracy and timing; Patient will grasp the pen like any writing tool with the thumb, index finger and middle finger. Patient will hold the pen at no less than a 45 angle from the writing space. An infra-red light and fiber optic sensor in the tip of the pen sense reflect as the user traces a pattern with the pen and provide immediate auditory feedback if the user wanders off the pattern.
eye hand coordination movement speed subjectively | baseline
  wall catch test will be used to assess eye hand coordination movement speed;A bucket of tennis balls will be available directly in front of the participant and a ball will be held in the dominant hand. The physical therapist will count down '3, 2, 1, go' and start the stopwatch, the ball will be thrown underarm off the wall and the return will be caught in their opposing hand. The participant then continue to throw and catch the ball in alternative hands for 30 s. If a ball is dropped, participants will be instructed to reach into the bucket of balls and to continue the test as quickly as possible.
eye hand coordination upper and limb muscles coordination | baseline
  standardized finger to nose test will be used to assess eye hand coordination upper and limb muscles coordination; Test will be performed with patient starting position then the patient will be asked to bring the tip of index finger to the tip of his nose then to touch a target 45 cm at arm's length and return to touch their nose again. It consists of recording how many times the individuals alternately touched their tip of their nose and a target placed in front of them on a wall